CLINICAL TRIAL: NCT05053269
Title: Association of Body Weight Growth After Birth and Bronchopulmonary Dysplasia(BPD)
Brief Title: Body Weight Growth After Birth and Bronchopulmonary Dysplasia
Status: Withdrawn | Type: Observational
Why Stopped: none was included
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 2020228
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-10

CONDITIONS: Bronchopulmonary Dysplasia; Preterm
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good body weight growth: body weight growth after birth is consistent with the growth curve
  Interventions: Other: good body weight growth
- poor body weight growth: body weight growth after birth is inconsistent with the growth curve
  Interventions: Other: poor body weight growth

INTERVENTIONS:
Other: good body weight growth — body weight growth after birth is consistent with the growth curve
  Groups: good body weight growth
Other: poor body weight growth — body weight growth after birth is inconsistent with the growth curve
  Groups: poor body weight growth

SUMMARY:
Bronchopulmonary dysplasia (BPD) is one of the most common, complex, and severe diseases in preterm infants. BPD was first described as chronic pulmonary disease in survivors of severe respiratory distress syndrome (RDS) in 1967, which was also called as the "old" BPD. In recent years, the definition for BPD has developed a lot. The National Institute of Child Health and Human Development (NICHD) workshop in 2018 assessed BPD at 36 post-menstrual age (PMA) along with radiographic confirmation and used a severity grading of I-III. Although with effective surfactant supplement and oxygen support, BPD brings a great challenge to neonatologists.

DETAILED DESCRIPTION:
Besides persistent inflammation, prolonged invasive ventilation and oxidative damage. body weight is the one of the most important factors to induce BPD. Poor extrauterine growth is commonly described in extremely preterm infants. But, the relationship of postnatal growth with BPD and respiratory morbidity is not entirely understood.

The aim of the present study is to assess whether body weight growth after birth is the risk factor for BPD.

ELIGIBILITY:
Inclusion Criteria:

* equal to or less than 32 weeks' gestational age

Exclusion Criteria:

* main congenital malformation
* parents' refusal

Ages: 1 Minute to 1 Day | Sex: All
Age Groups: Child
Study Population: the preterm infants' gestational age is equal to or less than 32 weeks will be included in the study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of BPD | up to 36 weeks' gestational age
  the infant was diagnosed with BPD

SECONDARY OUTCOMES:
body weight growth after birth | up to 36 weeks' gestational age
  to assess whether body weight growth after birth is consistent with the growth curve

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided